CLINICAL TRIAL: NCT00051207
Title: Interpersonal Psychotherapy for Depression With Co-occurring Panic and Anxiety Symptoms (IPT-PS)
Brief Title: Therapy for Depression With Co-occurring Panic or Anxiety Symptoms
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH061948 (NIH); DSIR AT-AS
Record Dates: First submitted 2003-01-07; First posted 2003-01-08 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2007-12

CONDITIONS: Depression; Anxiety Disorders; Panic Disorder
Keywords: Mood Disorders; Psychotherapy; Comorbidity
MeSH Terms: conditions — Depression; Anxiety Disorders; Panic Disorder; Mood Disorders | interventions — Interpersonal Psychotherapy; adenylate isopentenyltransferase

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy (IPT)
Behavioral: IPT for Depression with Co-occurring Panic and Anxiety Symptoms (IPT-PS)

SUMMARY:
This 6-month study, with a 3-month follow up period, will compare the effectiveness of new and traditional psychotherapies for depression with panic or anxiety symptoms.

DETAILED DESCRIPTION:
Many depressed patients also experience significant symptoms of panic or anxiety. This study will compare the effectiveness of a new therapy called interpersonal psychotherapy for depression with panic or anxiety symptoms (IPT-PS) with that of traditional interpersonal psychotherapy for depression (IPT).

Participants are randomly assigned to receive up to 24 weeks of treatment with either IPT-PS or traditional IPT. Improvements in interpersonal functioning, quality of life, and symptoms of depression and anxiety will be assessed at the end of therapy and at a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of major depression with co-existing panic or anxiety symptoms.

Exclusion Criteria:

* History of manic episode(s). Patients who have had hypomanic episodes in the past will be accepted into the study, provided they meet other admission criteria and are not presenting in a current hypomanic or mixed episode.
* History of schizophrenia or schizoaffective disorder.
* Organic affective syndrome.
* Unspecified functional psychosis.
* Anorexia nervosa or bulimia nervosa. Patients meeting criteria for an eating disorder not otherwise specified will not be excluded.
* Chronic drug or alcohol abuse/dependence within the past 2 years. Patients with abuse related to episodes will not be excluded.
* DSM-IV criteria for borderline or antisocial personality disorder. Patients who meet criteria for other Axis II disorders will not be excluded.
* Inpatient treatment due to suicide risk or psychotic symptoms.
* Index episode secondary to the effect of medically prescribed drugs.
* Significant or untreated medical illness, including cardiovascular disorder, renal or liver disease, epilepsy, untreated hypertension, or unstabilized endocrine disease.
* Medical illness that would interfere with the best treatment strategy for the potential participant.
* Current treatment with an antidepressant. Patients on a stable dose of anxiolytics for at least 3 months prior to study participation who are able to maintain this dosage throughout the study will not be excluded.
* Pregnant and breast-feeding women will be accepted into the study, but will not be prescribed adjunctive medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36
Dates: Start 2002-11; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Western Psychiatric Institute and Clinic - Depression and Manic Depression Program, Pittsburgh, Pennsylvania, United States